CLINICAL TRIAL: NCT04858815
Title: Using Yogic Breathing to Reduce Stress in Anesthesia Personnel As Measured by Hair Cortisol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105235
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Stress; Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: single arm longitudinal trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of yogic breathing program (Experimental): This will be a single arm longitudinal trial designed to evaluate the feasibility and estimate the efficacy of implementing a self-administered yogic breathing program for stress reduction among anesthesiology practitioners at one academic medical center.
  Interventions: Behavioral: yogic breathing

INTERVENTIONS:
Behavioral: yogic breathing — participation in yogic breathing

SUMMARY:
Mind body exercises have long been used as a way for individuals to reduce stress and improve well-being. Recent studies indicate that yogic breathing (YB, also known as pranayama) could potentially impact both the mind and body by engaging both the physiological and neural elements and can thus be a specific tool that can be utilized by healthcare workers to combat burnout and decrease perceived levels of stress. Our aim is to understand and measure both subjectively and objectively the effects of long-term yogic breathing on stress levels in anesthesia personnel. This will be a single arm longitudinal trial designed to evaluate the feasibility and estimate the efficacy of implementing a yogic breathing program for stress reduction among anesthesiology practitioners at one academic medical center. The primary aim of the trial is to estimate the correlation between participant stress with average duration of yogic breathing over time. Secondarily the feasibility of implementing yogic breathing practices among anesthesiology practitioners will be evaluated. Feasibility measures will include recruitment rates, retention at 1year follow-up, and adherence to the yogic breathing program at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All clinical members of the MUSC anesthesia department (Attending physicians, resident physicians, and CRNAs)

Exclusion Criteria:

* Pregnancy (or anticipated pregnancy)
* chronic steroid use
* inadequate hair length for testing (less than 3cm at the back of the head)
* residents with anticipated graduation within the next one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Correlation of participant stress with average duration of yogic breathing over time | baseline & 12 month visit
  The study will estimate the efficacy of self-administered yogic breathing on participant stress over time using (a) cortisol levels measured in hair and (b) using validated survey instruments estimated as the change in stress from baseline to 12 months. The primary measure of efficacy is correlation between cortisol/stress levels with average weekly duration of yogic breathing in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Grayce Davis, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States